CLINICAL TRIAL: NCT01415622
Title: Feasibility, Efficacy, and Safety of Venous Ulcer Treatment Using a Hand Plasma Generator (PlasmaDerm) Chronisch venöser Ulzerationen (PlasmaDerm)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cinogy GmbH (Industry)
Collaborators: Institut fuer anwendungsorientierte Forschung und klinische Studien GmbH (Other); University Medical Center Goettingen (Other)
Responsible Party: Dirk Wandke, Cinogy GmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20101028
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2011-08

CONDITIONS: Venous Insufficiency
Keywords: plasma therapy; ulcus cruris
MeSH Terms: conditions — Venous Insufficiency; Foot Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PlasmaDerm (Experimental): Treatment of small to medium-sized Ulcera crurum with the PlasmaDerm VU-2010 device in addition to standard care.
  Interventions: Device: PlasmaDerm
- standard care (Other): standard care of Ulcera crurum
  Interventions: Procedure: standard care of Ulcera crurum

INTERVENTIONS:
Device: PlasmaDerm — plasma treatment 3 times a week for 8 weeks, 45 sec / cm² of Ulcus cruris size, in addition to standard care.
  Arms: PlasmaDerm
Procedure: standard care of Ulcera crurum — standard care of Ulcera crurum: Mepithel gaze for non-exsudative wounds, Mepilex for exsudative wounds, followed by surgical hose treatment. Additionally, a standardized compression therapy with Ulcer X is applied.
  Arms: standard care

SUMMARY:
The purpose of this study is to prove the safety and efficacy of plasma as an add-on treatment in combination with conventional treatment in cases of chronical venous Ulcus cruris.

DETAILED DESCRIPTION:
Ulcus cruris consists of pathologically changed tissue of the lower leg. Up to 80% are of venous origin. Because of the high prevalence of up to 2% the treatment of Ulcus cruris is of special economical importance. Depending on the size, depth and possible infections, the conventional treatment of these wounds consists of an adequate compression, preparation of the lesion, cover and of appropriate control of infections. All tasks are undertaken in order to faciliate the healing of these chronic wounds.

Plasma consists of free ions or electrons and can be created by various techniques. Commonly, it is use in the sterilization of medicinal equipment, the cauterization of tissue and in the field of coagulation. Because of its bactericidal characteristics, the direct interaction of plasma created by temperatures below 40°C on tissue is intensively studied. Both in vitro and in vivo studies proved a significant reduction of bacterial contamination in different test systems. As bacterial contamination might slow down wound healing, plasma treatment might be a useful tool to complement conventional methods in the treatment of chronical wounds.

ELIGIBILITY:
Inclusion Criteria:

* persons of both gender aged 50 and older; females must be in menopause for at least one year
* at least one chronical venous ulcerisation at one or both legs with the following characteristics: size between 5 cm² and 30 cm²; duration 12 weeks to 10 years; located between knee and ankle; dermis and subkutis being involved, without damage of muscles, bones or tendon
* vital wound ground with granulation tissue
* proof of ulcerisation caused by venous malformation by duplex sonography, the tibiobrachiale index being between 0.8 and 1.3
* no active wound treatment one week before study treatment starts

Exclusion Criteria:

* females not being in menopause
* non-venous cause for ulzerisation
* lymphatic oedema, wound infection, necrotic tissue, venous fistula, bradytrophe wound ground
* clinical treatment of the venes during the last three months
* background therapy with systemic corticosteroides above Cushing-level (7.5 mg Prednisolonequivalent)
* previous radiation treatment of the ulzerisation area
* patients with defibrillator, after organ transplantation, cardiac insufficiency, known connective tissue disease, malnutrition (Albumin i.S. < 2.5 g/dl), Diabetes mellitus (HbA1c > 8%), active maligne disease, severe rheumatoide arthritis, hemodialysis, active sickle cell anemia
* known alcohol or drug abuse
* patients currently participating or having participated during the last 4 weeks in another clinical trial
* patients being unable to understand the intention of the clinical trial
* patients being not compliant or not being independant from the sponsor or investigator
* missing approval to collect and process pseudomized data
* hospitalization in a mental institution due to § 20 MPG

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
number of SAEs | 2 months

SECONDARY OUTCOMES:
inflammation of the Ulcus crurus | 2 months
size of the Ulcus crurus | once a week
pain assessment between treatments | 2 months
pain assessment during treatment | 2 months
patient satisfaction (patient-benefit-index) | 2 months
overall assessment of the treatment from patient's view | 2 months
overall assessment of the treatment from investigator's view | 2 months
relapse rate 4 weeks after end of treatment | after 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Emmert, Prof., Principal Investigator — Dept. of Dermatology, Venerology and Allergology, Göttingen University Hospital
Locations (1):
- Dep. of Dermatology, Venerology and Allergology, Göttingen University Hospital, Göttingen, Germany

REFERENCES:
- [Derived] Brehmer F, Haenssle HA, Daeschlein G, Ahmed R, Pfeiffer S, Gorlitz A, Simon D, Schon MP, Wandke D, Emmert S. Alleviation of chronic venous leg ulcers with a hand-held dielectric barrier discharge plasma generator (PlasmaDerm((R)) VU-2010): results of a monocentric, two-armed, open, prospective, randomized and controlled trial (NCT01415622). J Eur Acad Dermatol Venereol. 2015 Jan;29(1):148-55. doi: 10.1111/jdv.12490. Epub 2014 Mar 25. PMID 24666170
- See also: Related Info — http://www.cinogy.de/